CLINICAL TRIAL: NCT05171790
Title: A Multicenter, Open Phase 1b Study to Evaluate the Efficacy and Safety of QL1706 Injection in Patients With Advanced Malignant Solid Tumors
Brief Title: A Study to Evaluate the Efficacy and Safety of QL1706 Injection in Patients With Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QL1706-102
Record Dates: First submitted 2021-11-30; First posted 2021-12-29 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QL1706 injection (Experimental): This clinical trail is a single arm study, all the patients that meet the entry criteria will receive treatment until disease progression occurs or meet other criteria for the discontinuation of treatment. QL1706 will be administered by intravenous infusion, 5 mg/kg, Q3W.
  Interventions: Drug: QL1706 injection

INTERVENTIONS:
Drug: QL1706 injection — 5 mg/kg, IV, Q3w
  Other Names: PSB205 injection

SUMMARY:
This a multi-center, open-label, non-randomized phaseⅠb trail. The purpose of this study was to evaluate the efficacy and safety of QL1706 in patients with advanced solid tumors and to investigate the immunogenicity and pharmacokinetic characteristics of QL1706.

DETAILED DESCRIPTION:
The study was divided into screening/baseline, treatment and follow-up periods. Efficacy assessment and safety monitoring will be conducted throughout the study period.

Subjects will continue study treatment until disease progression occurs (unless the investigator believes there is a sustained clinical benefit) or other criteria for discontinuing study treatment are met, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Subjects participate voluntarily and sign informed consent.
* Patients with Pathologically confirmed metastatic or recurrent malignant solid tumors，such as lung cancer, nasopharyngeal carcinoma, cervical cancer, hepatocellular carcinoma, kidney cancer etc., failure or intolerance of at least first-line treatment and unsuitable for radical treatment such as surgery
* Subject has at least one measurable lesion according to RECIST (V1.1) evaluation criteria.
* Eastern Cooperative Oncology Group (ECOG) score was 0 or 1.
* The extension of life is more than 3 months
* Vital organs' function is adequate for enrolling
* Subjects agree to use effective contraceptive measures.Women who have not been pregnant or breastfeeding.
* Before the first use of the investigational drug, all the reversible toxicity of the previous antitumor therapy returned to ≤1 (according to CTCAE V5.0),Excluding any grade of hair loss and pigmentation, grade 2 or less peripheral sensory neuropathy, and other abnormalities that the investigator and/or sponsor assessed to outweigh the risk of toxicity.

Exclusion Criteria:

* Active autoimmune diseases that exist within 2 years prior to the first use of the investigational drug and require systemic treatment.
* There are known past grade 3 or 4 immune-related adverse events associated with antitumor immunotherapy.
* Symptomatic central nervous system (CNS) metastasis, pia metastasis or spinal cord compression due to metastasis prior to signing informed consent.
* Subjects with any of the following cardiovascular diseases that seriously endanger the safety of the subjects or affect the completion of the study
* Subjects with diseases that are planned to be treated with systemic corticosteroids or other immunosuppressive drugs during the study period
* Prior treatment with cytotoxic T lymphocyte-associated antigen-4 (CTLA-4) inhibitor combined with programmed cell death protein-1 (PD-1) inhibitor, or CTLA-4 inhibitor combined with PD-L1 inhibitor.
* Had received chemotherapy, targeted therapy, biotherapy, endocrine therapy, immunotherapy and other anti-tumor treatments within 4 weeks before the first use of experimental drugs
* Subjects with positive antibodies to HIV;Treponema pallidum antibody positive;HBsAg positive patients with VIRAL DEoxy ribonucleic acid (HBV DNA) >2000 IU/ mL or 10^4 copy number/mL should receive antiviral therapy according to local treatment guidelines and be willing to receive antiviral therapy throughout the study period.Hepatitis C virus antibody positive and viral ribonucleic acid (HCV RNA) positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 419 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
objective response rate (ORR) | up to 24 weeks
  ORR includes complete response (CR) and partial response (PR) cases. According to RECIST V1.1, the first appearance of PR or CR requires additional imaging to confirm the lesion at ≥4 weeks.

SECONDARY OUTCOMES:
disease control rate (DCR) | up to 24 weeks
  DCR refers to the percentage of the cases in which the best efficacy rating is complete response (CR) or partial response (PR) or stable disease (SD).
progression-free survival (PFS) | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Progression-free survival (PFS) is defined as the time between a subject's first infusion QL1706 injection and their first radiographic evaluation of disease progression or death from any cause, whichever comes first.
overall survival time (OS) | From date of enrollment until the date of death from any cause, assessed up to 24 months
  Overall survival (OS) is the time between the subject's first infusion QL1706 injection and death from any cause.
adverse event (AE) | up to 90 days after the last QL1706 injection is administered.
  The rates and severity of AEs after QL1706 injection

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, Doctor, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ma Y, Lin S, Chen Q, Xue J, Yang Y, Zang A, Cheng Y, Zhang Y, Wang X, Chen Z, Qu S, He J, Chen C, Jin C, Zhu D, Li Q, Liu X, Su W, Ba Y, Li W, Li Q, Zhu C, Huang Z, Kang X, Xue S, Li H, Wang C, Luo F, Huang Y, Zhang L, Zhao H. Updated efficacy and predictive biomarkers of QL1706, a bifunctional PD-1/CTLA-4 dual blocker in advanced solid tumors-A phase 1/1b study. Cell Rep Med. 2025 Oct 21;6(10):102396. doi: 10.1016/j.xcrm.2025.102396. Epub 2025 Oct 3. PMID 41045933
- [Derived] Zhao Y, Ma Y, Zang A, Cheng Y, Zhang Y, Wang X, Chen Z, Qu S, He J, Chen C, Jin C, Zhu D, Li Q, Liu X, Su W, Ba Y, Hao Y, Chen J, Zhang G, Qu S, Li Y, Feng W, Yang M, Liu B, Ouyang W, Liang J, Yu Z, Kang X, Xue S, Yang G, Yan W, Yang Y, Liu Z, Peng Y, Fanslow B, Huang X, Zhang L, Zhao H. First-in-human phase I/Ib study of QL1706 (PSB205), a bifunctional PD1/CTLA4 dual blocker, in patients with advanced solid tumors. J Hematol Oncol. 2023 May 8;16(1):50. doi: 10.1186/s13045-023-01445-1. PMID 37158938